CLINICAL TRIAL: NCT00604201
Title: Co-Infusion of Umbilical Cord Blood and Haploidentical CD34+ Cells Following Nonmyeloablative Conditioning as Treatment for Severe Aplastic Anemia and MDS Associated With Severe Neutropenia Refractory to Immunosuppressive Therapy
Brief Title: Stem Cell Transplant Using Peripheral and Cord Blood Stem Cells to Treat Severe Aplastic Anemia and Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080046; 08-H-0046; NCT00608413 (obsolete NCT alias)
Record Dates: First submitted 2008-01-08; First posted 2008-01-30 (Estimated); Results first posted 2020-07-31 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Myelodysplastic Syndrome (MDS) With Refractory Anemia (RA); Severe Aplastic Anemia (SAA)
Keywords: Nonmyeloablative; Haploidentical; Umbilical Cord Blood; SAA; Severe Aplastic Anemia; Myelodysplastic Syndrome; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Aplastic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Co-infusion of UCB and Haploidentical CD34+ cells (Experimental): Stem cell recipients received co-infusion of unrelated umbilical cord blood (UCB) and haploidentical CD34+ cells from a related donor following non-myeloablative conditioning for neutropenic patients with severe aplastic anemia (SAA) or myelodysplastic syndrome (MDS) with refractory anemia (RA)
  Interventions: Biological: Umbilical Cord Blood

INTERVENTIONS:
Biological: Umbilical Cord Blood — unrelated umbilical cord blood will be co-infused with haploidentical CD34-selected cells from a related donor for treatment of severe aplastic anemia and myelodysplastic syndrome.

SUMMARY:
This study will evaluate the safety and effectiveness of treating patients with severe aplastic anemia (SAA) or myelodysplastic syndrome (MDS) with both peripheral blood stem cells from a family member and umbilical cord blood stem cells from an unrelated donor.

Patients with SAA or MDS for whom other treatments have failed or are not available may be eligible for this study. Candidates may not have a tissue-matched sibling or matched unrelated donor and must have a family member who is a partial tissue type match.

Participants undergo the following tests and procedures:

* Insertion of a central intravenous (IV) line (plastic tube) into a large vein. The tube is used for giving the donated stem cells and antibiotics and other medicines, for transfusions of red blood cells and platelets, and for collecting blood samples.
* Preparatory chemotherapy (fludarabine, cyclophosphamide and anti-thymocyte globulin) and total body irradiation to suppress immunity and prevent rejection of the donated cells.
* Infusion of the donated stem cells and umbilical cord cells.
* Immune suppression with the drugs tacrolimus, mycophenolate mofetil and prednisone to prevent rejection of the donated cells and to prevent graft-versus-host disease (GVHD), a complication of stem cell transplants in which the donors immune cells destroy the patients healthy tissues.

The average hospital stay after stem cell transplantation is 3 to 4 weeks. Patients return for frequent follow-up visits for the first 2 to 4 months after transplantation. Once the patient returns home, his or her referring physician is asked to send results of any laboratory testing to the NIH researchers at least every 3 months for the first 3 years and annually thereafter. Patient follow-up visits are scheduled at NIH at 1, 2, 3, 4 and 5 years after transplantation to monitor for signs of disease or post-transplantation complications, such as infection or GVHD. After 5 years, participants are offered the opportunity to enroll in NHLBIs long-term evaluation and follow-up care protocol.

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA) and myelodysplastic syndrome (MDS) are life-threatening bone marrow disorders. For SAA patients, long term survival can be achieved with immunosuppressive treatment. However, of those patients treated with immunosuppressive therapy, one quarter to one third will not respond, and about 50 percent of responders will relapse.

Allogeneic bone marrow transplantation from either HLA-matched sibling or matched unrelated donor cures about 70 percent of patients with SAA and 30-60 percent of patients with MDS. Unfortunately, most patients with these disorders are not suitable candidates for hematopoietic stem cell transplantation (HSCT) due to advanced age or lack of a histocompatible donor. For such patients, transplantation using unrelated cord blood (UCB) has been shown to be a reasonable alternative transplant strategy. The advantage to UCB transplant is the ease and rapidity of availability, requirement of less than perfect HLA match, and lower rates of graft versus host disease compared to mismatched bone marrow or peripheral blood stem cell transplants. The major disadvantage of UCB transplantation in adults is the limited number of nucleated cells contained within the cord unit resulting in prolonged neutropenia and failure of engraftment which contributes to infection and transplant related mortality (TRM). In order to harness the advantage of UCB availability and to overcome the disadvantage of delayed neutrophil recovery, we propose to test whether co-administration of unrelated umbilical cord blood and a relatively low number of highly purified haploidentical peripheral blood CD34+ cells from a related donor might promote rapid engraftment and reduce TRM secondary to prolonged neutropenia associated with conventional umbilical cord blood transplant (UCBT).

This research protocol is therefore designed to evaluate the safety and effectiveness of co-infusion of unrelated umbilical cord blood and haploidentical CD34 plus cells from a related donor following nonmyeloablative conditioning for neutropenic patients with SAA or MDS with refractory anemia (RA) that has proven to be refractory to medical therapy. Subjects will receive a novel non-myeloablative immunosuppressive conditioning regimen of cyclophosphamide, fludarabine, horse ATG (antithymocyte globulin) and one dose of total body irradiation (200cGy) followed by an infusion of the allografts. The haploidentical stem cell product will be T-cell depleted and enriched for CD34 plus cells using the Miltenyi CliniMacs system. To reduce TRM secondary to prolonged neutropenia associated with conventional UCB transplantation, haploidentical CD34+ stem cells will be co-infused with a single UCB unit (serologically matched at greater than or equal to 4/6 HLA loci).

The primary endpoint is donor engraftment by day 42 (defined as an ANC of greater than 500 from either the haplo donor, the cord, or both combined). Secondary endpoints will include standard transplant outcome variables such as non-hematological toxicities, incidence and severity of acute and chronic GVHD, and relapse of disease. We will also evaluate ANC recovery (ANC greater than 500 cells/microl) at day 22, and 100 day and 200 day treatment related mortality (TRM) of this novel transplant approach. Health related quality of life will also be assessed pre-transplant 30 and 100 days post-transplant, and every 6 months until 5 years post transplant.

ELIGIBILITY:
* INCLUSION CRITERIA - RECIPIENT:
* Diagnosed with severe aplastic anemia characterized by all of the following:

  1. Bone marrow cellularity less than 30 percent (excluding lymphocytes)
  2. Transfusion dependence for platelets and/or red blood cells (RBCs)
  3. Neutropenia (absolute neutrophil count less than 500 cells/microL) OR for patients receiving granulocyte transfusions, absolute neutrophil count < 500 cells/microL before beginning granulocyte transfusions].)

OR

* Diagnosed with myelodysplastic syndrome characterized by refractory anemia OR refractory anemia with ringed sideroblasts (RARS and at least one of the following:

  1. Neutropenia [(absolute neutrophil count < 500 cells/microL) OR for patients receiving granulocyte transfusions, absolute neutrophil count < 500 cells/microL before beginning granulocyte transfusions]) and history of 1 or more opportunistic infections related to neutropenia. OR
  2. History of severe aplastic anemia transformed to MDS
* Intolerance of or failure to respond standard immunosuppressive therapy.
* Availability of at least one HLA-haploidentical (i.e. greater than or equal to 5/10 and less than or equal to 8/10 HLA match) related donor (HLA-A, B, C, DR, and DO loci) who is available to donate CD34+ cells (4-75 years old).
* Availability of at least one 4/6 HLA-matched (HLA-A, B, and DR loci) cord blood unit from the National Marrow Donor Program (NMDP). The cord blood unit must contain a minimum total nucleated cells (TNC) (prior to thawing) of at least 1.5 x 10(7) cells per kilogram of recipient body weight with the following exception: if the minimum criterion of TNC is not met the cord unit must contain at least 1.7 x 10(5) CD34 plus cells/kg (prior to thawing).
* Ages 4-55 years inclusive.
* Ability to comprehend the investigational nature of the study and provide informed consent. The procedure will be explained to subjects aged 4-17 years with formal consent being obtained from parents or legal guardian.

  * Telomere Length Testing
  * In patients where a suspicion for a familial bone marrow failure syndromes (BMFS) exists, TERC and TERT mutation testing will be performed on protocol 04-H-0012 or performed elsewhere prior to enrolling on 04-H-0012.

EXCLUSION CRITERIA - RECIPIENT:

* Availability of an HLA identical or 9/10 HLA matched(HLA A, B, C, DR, and DO loci-relative to serve as a stem cell donor.
* The patient is deemed to be a candidate for a 6/6 HLA matched unrelated stem cell transplant (availability of a donor and resources required for such a transplant).
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or more.
* Major anticipated illness or organ failure incompatible with survival from transplant
* Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the transplant treatment unlikely and making informed consent impossible.
* Positive pregnancy test for women of childbearing age.
* HIV positive
* Diagnosis of Fanconi anemia (by chromosome breakage study).
* Diffusion capacity of carbon monoxide (DLCO) less than 40 percent using DLCO corrected for Hgb or lung volumes (patients under the age of 10 may be excluded from this criterion if they have difficulty performing the test correctly and thus are unable to have their DLCO assessed) using DL Adj and DL/VA/Adj.
* Left ventricular ejection fraction less than 40 percent (evaluated by ECHO)
* Transaminases greater than 5x upper limit of normal (when transaminases are elevated, the subject may be excluded at the discretion of the PI).
* Serum bilirubin greater than 4 mg/dl
* Creatinine clearance less than 50 cc/min by 24 hr urine collection (adjusted for body surface area, i.e.50 ml/min/1.73m(2))
* Serum creatinine > 2.5 mg/dl
* Failure to collect an adequate number of CD34+ cells (i.e. greater than or equal 2 x 10(6) CD34+ cells/kg) for transplantation from the subject s haploidentical relative.
* Presence of an active infection not adequately responding to appropriate therapy
* History of a malignant disease liable to relapse or progress within 5 years

INCLUSION CRITERIA - RELATED HAPLOIDENTICAL DONOR DONATING PURIFIED CD34 PLUS CELLS:

* HLA mismatched family donor (greater than or equal to 5/10 and less than or equal to 8/10 HLA matched (HLA-A, B, C, DR and DO loci) who is available to donate CD34+ cells.
* Ages 4-75 inclusive
* Weight greater than or equal to 15 kg.
* For adults: Ability to comprehend the investigational nature of the study and provide informed consent. For minors: Written informed consent from one parent or guardian who is not the recipient of the transplant and informed assent: The process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.
* If there is a suspicion of familial BMFS in the recipient, then the donor must have undergone genetic testing for genes associated with BMFS - performed at a CLIA-certified laboratory, prior to enrolling in this protocol.

EXCLUSION CRITERIA RELATED DONOR (ANY OF THE FOLLOWING):

* Pregnant or breastfeeding.
* A suitable adult haplo identical donor is available.
* Unfit to receive filgrastim (G-CSF) and undergo apheresis (history of stroke, MI, unstable angina, uncontrolled hypertension, severe heart disease or palpable spleen).
* HIV positive (Donors who are positive for HBV, HCV or HTLV I/II, T. cruzi [Chagas] may be used at the discretion of the investigator following counseling and approval from the recipient).
* Sickling hemoglobinopathies including HbSS, HbAS, HbSC. Donors with HbAS are acceptable.
* Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the BMT treatment unlikely and making informed consent impossible.
* Screening test positive for Chagas disease (Trypanosoma cruzi /T. cruzi/trypanosomiasis) confirmed by the Center for Disease Control (CDC).

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-05-21 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2021-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Childs, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Young NS, Barrett AJ. The treatment of severe acquired aplastic anemia. Blood. 1995 Jun 15;85(12):3367-77. No abstract available. PMID 7780125
- [Background] Young NS, Maciejewski J. The pathophysiology of acquired aplastic anemia. N Engl J Med. 1997 May 8;336(19):1365-72. doi: 10.1056/NEJM199705083361906. No abstract available. PMID 9134878
- [Background] Zoumbos NC, Gascon P, Djeu JY, Trost SR, Young NS. Circulating activated suppressor T lymphocytes in aplastic anemia. N Engl J Med. 1985 Jan 31;312(5):257-65. doi: 10.1056/NEJM198501313120501. PMID 2981406
- [Derived] Giudice V, Wu Z, Kajigaya S, Fernandez Ibanez MDP, Rios O, Cheung F, Ito S, Young NS. Circulating S100A8 and S100A9 protein levels in plasma of patients with acquired aplastic anemia and myelodysplastic syndromes. Cytokine. 2019 Jan;113:462-465. doi: 10.1016/j.cyto.2018.06.025. Epub 2018 Jun 27. PMID 29958797
- [Derived] Giudice V, Banaszak LG, Gutierrez-Rodrigues F, Kajigaya S, Panjwani R, Ibanez MDPF, Rios O, Bleck CK, Stempinski ES, Raffo DQ, Townsley DM, Young NS. Circulating exosomal microRNAs in acquired aplastic anemia and myelodysplastic syndromes. Haematologica. 2018 Jul;103(7):1150-1159. doi: 10.3324/haematol.2017.182824. Epub 2018 Apr 19. PMID 29674506
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-H-0046.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
Started | 31
Completed | 21
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 4
  More than one race | 4
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Who Developed Chronic GVHD
Description: Participants who developed chronic graft-versus-host disease (GVHD)
Time Frame: 5 years
Population: All recipients that received unrelated umbilical cord blood (UCB) and haploidentical CD34+ cells
Measure: Count of Participants; unit: Participants
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
Number analyzed (Participants) | 31
Participants | 12

2. Secondary Outcome: Number of Participants Who Developed Acute GVHD
Description: Participants who had acute graft-versus-host disease (GVHD)
Time Frame: 100 days
Population: All recipients that received unrelated umbilical cord blood (UCB) and haploidentical CD34+ cells
Measure: Count of Participants; unit: Participants
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
Number analyzed (Participants) | 31
Participants | 5

3. Primary Outcome: Number of Participants Who Engrafted by Day 42
Description: Participants who reached engraftment by day 42 (±3 days) defined as an absolute neutrophil count (ANC) of U> U500 cells/µl
Time Frame: 42 days
Population: All recipients that received unrelated umbilical cord blood (UCB) and haploidentical CD34+ cells
Measure: Count of Participants; unit: Participants
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
Number analyzed (Participants) | 31
Participants | 30

4. Secondary Outcome: Number of Participants Who Experienced Treatment Related Mortality (TRM) Day 100
Description: Number of participants who experienced treatment related mortality (TRM) by day 100
Time Frame: 100 days
Population: All recipients that received unrelated umbilical cord blood (UCB) and haploidentical CD34+ cells
Measure: Count of Participants; unit: Participants
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
Number analyzed (Participants) | 31
Participants | 1

5. Secondary Outcome: Number of Participants Who Experienced Treatment Related Mortality (TRM) Day 200
Description: Number of participants who experienced treatment related mortality (TRM) by day 200
Time Frame: 200 days
Population: All recipients that received unrelated umbilical cord blood (UCB) and haploidentical CD34+ cells
Measure: Count of Participants; unit: Participants
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
Number analyzed (Participants) | 31
Participants | 1

6. Secondary Outcome: Number of Participants Who Had ANC Recovery at Day 22
Description: Number of participants who reached engraftment by day 22 (±3 days) defined as an ANC of U> U500 cells/µl
Time Frame: 22 days
Population: All recipients that received unrelated umbilical cord blood (UCB) and haploidentical CD34+ cells
Measure: Count of Participants; unit: Participants
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
Number analyzed (Participants) | 31
Participants | 30

7. Secondary Outcome: Number of Participants Who Had Relapse of Disease
Description: Participants who had experienced relapse of disease
Time Frame: 5 years
Population: All recipients that received unrelated umbilical cord blood (UCB) and haploidentical CD34+ cells
Measure: Count of Participants; unit: Participants
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
Number analyzed (Participants) | 31
Participants | 1

8. Secondary Outcome: Number of Participants Who Developed Grade II Acute GVHD
Description: Participants who developed Grade II Acute GVHD as defined by CIMBTR criteria for Organ Stages of Acute GVHD.
  Stage II Acute GVHD: Skin - rash on 25-50 percent body surface area; Liver - Total Bilirubin 3.1-6.0 mg/dL; Lower GI - Diarrhea 1001-1500 mL/day.
  Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: 100 days
Population: All recipients that received unrelated umbilical cord blood (UCB) and haploidentical CD34+ cells
Measure: Count of Participants; unit: Participants
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
Number analyzed (Participants) | 31
Participants | 3

9. Secondary Outcome: Number of Participants Who Developed Grade III Acute GVHD
Description: Participants who developed Grade III Acute GVHD as defined by CIMBTR criteria for Organ Stages of Acute GVHD.
  Stage III Acute GVHD: Skin - Rash on >50% of body surface; Liver - Total Bilirubin 6.1 - 15.0 mg/dL; Lower GI - Diarrhea > 1500 mL/day
  Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: 100 days
Population: All recipients that received unrelated umbilical cord blood (UCB) and haploidentical CD34+ cells
Measure: Count of Participants; unit: Participants
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
Number analyzed (Participants) | 31
Participants | 2

10. Secondary Outcome: Number of Participants Who Developed Mild Chronic GVHD
Description: Participants who developed mild chronic graft vs host disease (GVHD).
  Mild chronic GVHD is 2 or fewer organs with no more than score 1 and no lung involvement. Mild disease is associated with a good prognosis whereas severe disease is associated with higher treatment-related mortality and lower survival.
  Organs are scored on a 0 to 3 scale from no involvement/no symptoms to severe functional compromise.
Time Frame: 5 years
Population: All recipients that received unrelated umbilical cord blood (UCB) and haploidentical CD34+ cells
Measure: Count of Participants; unit: Participants
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
Number analyzed (Participants) | 31
Participants | 10

11. Secondary Outcome: Number of Participants Who Developed Moderate Chronic GVHD
Description: Participants who experienced moderate chronic GVHD.
  Moderate GVHD is 3 or more organs with score 1, any organ with score 2, or lung with score 1, and usually requires systemic immune-suppressive treatment. Mild disease is associated with a good prognosis whereas severe disease is associated with higher treatment-related mortality and lower survival.
  Organs are scored on a 0 to 3 scale from no involvement/no symptoms to severe functional compromise.
Time Frame: 5 years
Population: All recipients that received unrelated umbilical cord blood (UCB) and haploidentical CD34+ cells
Measure: Count of Participants; unit: Participants
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
Number analyzed (Participants) | 31
Participants | 2

12. Secondary Outcome: Number of Participants Who Developed Severe Chronic GVHD
Description: Participants who developed severe chronic GVHD.
  Severe chronic GVHD is any organ with a score of 3 or lung with a score of 2, and means that substantial organ damage already exists. Mild disease is associated with a good prognosis whereas severe disease is associated with higher treatment-related mortality and lower survival
  Organs are scored on a 0 to 3 scale from no involvement/no symptoms to severe functional compromise.
Time Frame: 5 years
Population: All recipients that received unrelated umbilical cord blood (UCB) and haploidentical CD34+ cells
Measure: Count of Participants; unit: Participants
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
Number analyzed (Participants) | 31
Participants | 0

13. Secondary Outcome: Number of Participants Who Developed Steroid Refractory Acute GVHD
Description: Participants who had developed steroid refractory (not responding to standard steroid therapy) acute GVHD.
Time Frame: 100 days
Population: All recipients that received unrelated umbilical cord blood (UCB) and haploidentical CD34+ cells
Measure: Count of Participants; unit: Participants
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
Number analyzed (Participants) | 31
Participants | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Co-infusion of UCB and Haploidentical CD34+ Cells
All-Cause Mortality (participants affected / at risk) | 5/31
Serious Adverse Events (participants affected / at risk) | 28/31
Other Adverse Events (participants affected / at risk) | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-infusion of UCB and Haploidentical CD34+ Cells (N=31)
Epstein-Barr virus associated lymphoproliferative disorder (Blood and lymphatic system disorders) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (7)
Haemolysis (Blood and lymphatic system disorders) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Systolic dysfunction (Cardiac disorders) | 2 (2)
Ear infection (Ear and labyrinth disorders) | 1 (1)
Hyperglycaemia (Endocrine disorders) | 1 (1)
Scleritis (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Acute graft versus host disease in intestine (Gastrointestinal disorders) | 2 (3)
Chronic graft versus host disease in intestine (Gastrointestinal disorders) | 2 (2)
Clostridium difficile colitis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 1 (3)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Adverse drug reaction (General disorders) | 3 (4)
Acute graft versus host disease in intestine (Immune system disorders) | 1 (1)
Acute graft versus host disease in liver (Immune system disorders) | 1 (1)
Acute graft versus host disease in skin (Immune system disorders) | 1 (1)
Chronic graft versus host disease in skin (Immune system disorders) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (4)
Bacterial infection (Infections and infestations) | 1 (1)
BK virus infection (Infections and infestations) | 1 (2)
Capnocytophaga infection (Infections and infestations) | 1 (1)
Infection Reactivation, Cytomegalovirus infection (Infections and infestations) | 9 (21)
Encephalitis viral (Infections and infestations) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 2 (2)
Fungal skin infection (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Herpes virus infection (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 3 (4)
Metapneumovirus infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (2)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Posterior reversible encephalopathy syndrome (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Toxoplasmosis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Varicella zoster virus infection (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 3 (3)
Blood culture positive (Investigations) | 1 (1)
Body temperature increased (Investigations) | 7 (10)
Coronavirus test positive (Investigations) | 1 (1)
Stenotrophomonas test positive (Investigations) | 1 (1)
Urine electrolytes decreased (Investigations) | 1 (1)
Myotonia (Musculoskeletal and connective tissue disorders) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 3 (3)
Seizure (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal injury (Surgical and medical procedures) | 1 (1)
Dialysis device insertion (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT00604201/Prot_SAP_000.pdf